CLINICAL TRIAL: NCT04573790
Title: A Modified Rabbit Training Model for Establishing an Emergency Front of Neck Airway in Children
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: eFONA KISPI
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Emergency Front of Neck Airway in Children
Keywords: Cannot intubate, cannot oxygenate in children; emergency front of neck airway; rabbit cadaver model; emergency tracheotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trained in eFONA: Trained participants completed our eFONA workshop within the last six month prior to participating in this study
  Interventions: Procedure: eFONA
- Untrained in eFONA: Untrained participants had never taken part in our institutional eFONA workshop
  Interventions: Procedure: eFONA

INTERVENTIONS:
Procedure: eFONA — Surgical Tracheotomy

SUMMARY:
A "cannot intubate, cannot oxygenate" (CICO) situation is rare in paediatric anaesthesia, but can always occur in children under certain emergency situations. There is a paucity of literature on specific procedures for securing an emergency invasive airway in children under the age of 6 years. A modified emergency Front Of Neck Access (eFONA) technique using a rabbit cadaver model was developed to teach invasive airway protection in a CICO situation in children.

After watching an instructional video of our eFONA technique (tracheotomy, initial intubation with Frova catheter over which an endotracheal tube is inserted), 29 anaesthesiologists will perform two separate attempts on rabbit cadavers. The primary outcome is the success rate and the performance time overall and in subgroups of trained and untrained participants.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists working at the department of Anesthesia at University Children's Hospital Zurich

Exclusion Criteria:

* n.a.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiologists working at the department of Anesthesia at University Children's Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Sucess rate | during study period, approx 15min
  Correct positioning of the endotracheal tube in to the trachea
Performance time | during study period, max 240 sec
  Time needed to complete the surgical tracheotomy

SECONDARY OUTCOMES:
Secondary injuries | during study period, approx 15min
  paratracheal placement of the ETT, perforation of the back wall or complete rupture of the trachea

CONTACTS AND LOCATIONS:
Locations (1):
- University Childrens Hospital, Department of Anaesthesia and Children's Research Centre, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No